CLINICAL TRIAL: NCT02584660
Title: MulticEnter Trial of Rivaroxaban for Early disCharge of pUlmonaRY Embolism From the Emergency Department
Brief Title: A Study of Rivaroxaban for Early Discharge of Low Risk Pulmonary Embolism From the Emergency Department
Acronym: MERCURY PE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR107694; 39039039APE4001 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2015-09-11; First posted 2015-10-22 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Embolism
Keywords: Rivaroxaban; JNJ39039039; Pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Rivaroxaban; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Experimental): Participants will receive Rivaroxaban 15 milligram (mg) orally twice daily with food for the first 21 days followed by 20 mg orally once daily with food, for approximately 69 days for a total treatment duration of 90 days.
  Interventions: Drug: Rivaroxaban
- local Standard-of-care (Experimental): Participants will receive local Standard-of-care as per local protocol and defined by the medical team caring for the participant.
  Interventions: Drug: Standard-of-care

INTERVENTIONS:
Drug: Rivaroxaban — Participants will receive Rivaroxaban 15 milligram (mg) twice daily up to Days 21 by orally and Rivaroxaban 20 mg once daily up to Days 90 by orally.
  Arms: Rivaroxaban
Drug: Standard-of-care — Standard-of-care as per local protocol and defined by the medical team caring for the participant.
  Arms: local Standard-of-care

SUMMARY:
The purpose of the study is to evaluate that low risk Pulmonary Embolism (PE) participants who are discharged from the Emergency Department (ED) to the home environment and treated with rivaroxaban as outpatients have fewer total days in the hospital for bleeding and/or venous thromboembolism (VTE) events through Day 30 compared to participants who are treated with initial hospitalization and standard-of-care.

DETAILED DESCRIPTION:
This is a randomized (study medication is assigned by chance), open-label (all people know the identity of the intervention), parallel-group, multicenter (study conducted at multiple sites) study to evaluate that low risk PE participants who are discharged from the ED and treated with rivaroxaban compared to participants who are treated with initial hospitalization and standard-of-care. The study consists of a Screening and Randomization Period, followed by a 90-day open-label treatment period, and an end of study/early withdrawal (EOS) visit. The duration of study participation for each participant is approximately 3 months. The participants will be randomized in a 1:1 ratio to one of two treatments. Safety will be monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed acute symptomatic Pulmonary Embolism (PE) with or without symptomatic deep vein thrombosis (DVT)
* A PE participant diagnosed in the Emergency Department (ED) who is deemed to be at low risk of clinical deterioration as determined by the Hestia criteria
* Have no contraindications to and be able to complete randomized treatment and all study assessments
* Have a life expectancy of at least 6 months
* Must be willing and able to adhere to the prohibitions and restrictions specified in this protocol

Exclusion Criteria:

* Having received any Combined P-gp (P-glycoprotein) and strong CYP3A4 (Cytochrome P450) inhibitors (such as but not limited to ketoconazole, telithromycin or protease inhibitors) use within 4 days before randomization, or planned use during the study. Itraconazole use within 7 days before randomization or planned use during the study
* Having received any Combined P-gp and strong CYP3A4 inducers (such as but not limited to rifampin/rifampicin, rifabutin, rifapentine, phenytoin, phenobarbital, carbamazepine, or St. John's Wort) use within 2 weeks before randomization or planned use during the study
* Who Has contraindications to the use of any anticoagulant therapy (example, bleeding diathesis, history of gastrointestinal bleeding within 1 year or coagulopathy documented at Screening)
* Who Has known allergies, hypersensitivity, or intolerance to rivaroxaban or its excipients
* Woman who is pregnant, or breast-feeding, or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (50):
- United States (50):
  - Montgomery, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Los Angeles, California
  - Sacramento, California
  - Sylmar, California
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Pensacola, Florida
  - Tampa, Florida
  - Davenport, Iowa
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Jackson, Michigan
  - Lansing, Michigan
  - Royal Oak, Michigan
  - St Louis, Missouri
  - Atlantic City, New Jersey
  - Camden, New Jersey
  - Brooklyn, New York
  - Buffalo, New York
  - New York, New York
  - Stony Brook, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Toledo, Ohio
  - Zanesville, Ohio
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Bethlehem, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - West Reading, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Bellingham, Washington
  - Everett, Washington
  - Spokane, Washington
  - Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 300 participants screened, 114 participants were randomized (51 to rivaroxaban group and 63 participants in the standard-of-care group) and 112 participants were treated and received at least 1 dose of study agent.
Groups:
- Rivaroxaban: Participants received rivaroxaban 15 milligram (mg) twice daily up to Day 21 orally followed by rivaroxaban 20 mg once daily up to Days 90 orally.
- Standard-of-care: Participants received local Standard-of-care as per local protocol and is defined by the medical team caring for participants.
Period: Overall Study
Arm/Group | Rivaroxaban | Standard-of-care
Started | 51 | 63
Treated | 49 | 63
Completed | 44 | 55
Not Completed | 7 | 8
Not completed — Adverse Event | 4 | 0
Not completed — Lost to Follow-up | 3 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban | Standard-of-care | Total
Number analyzed (Participants) | 51 | 63 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (13.27) | 47.6 (17.22) | 48.3 (15.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 32 | 59
  Male | 24 | 31 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 47 | 60 | 107
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 14 | 34
  White | 29 | 48 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black or African American | 20 | 14 | 34
  Hispanic or Latino | 2 | 2 | 4
  Other | 1 | 1 | 2
  White | 29 | 48 | 77
  Not Hispanic or Latino | 47 | 60 | 107
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 51 | 63 | 114

OUTCOME MEASURES:

1. Primary Outcome: Mean Duration of Hospitalization
Description: Mean number of days of initial inpatient hospitalization (beginning from randomization to discharge from the hospital) plus any subsequent hospitalization(s) related to bleeding and/or venous thromboembolism (VTE) events up to 30 days were calculated.
Time Frame: Up to Day 30
Population: The intention to treat analysis set (ITT) included all participants who were randomized into the study.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Rivaroxaban | Standard-of-care
Number analyzed (Participants) | 51 | 63
Days | 0.191 (0.6862) | 1.393 (1.9642)
Statistical Analysis 1: Comparison: Rivaroxaban vs Standard-of-care; Test type: Superiority; p < .0001, t-test; Mean difference = -1.202, 95% CI 2-sided [-1.730 to -0.674]

2. Secondary Outcome: Percentage of Participants With Reoccurrence of Symptomatic Venous Thromboembolism Event (VTE) (Composite of Recurrent PE, New or Recurrent DVT) or VTE-related Death
Description: Reoccurrence of symptomatic, objectively confirmed VTE, defined as recurrent pulmonary embolism (PE) or new or recurrent deep vein thrombosis (DVT) (including symptomatic upper extremity DVT) or VTE related death were analyzed.
Time Frame: Up to 7, 14, 30, and 90 Days
Population: The ITT included all participants who were randomized into the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban | Standard-of-care
Number analyzed (Participants) | 51 | 63
Percentage of participants
  Up to 7 Days | 0 | 0
  Up to 14 Days | 0 | 0
  Up to 30 Days | 0 | 0
  Up to 90 Days | 0 | 0

3. Secondary Outcome: Percentage of Participants With Number of Unplanned Hospital Visits or Physician Office for VTE Symptoms and/or Bleeding
Description: Percentage of participants of unplanned hospitalization for VTE symptoms or bleeding-related hospital or physician visits were analyzed.
Time Frame: Up to 7, 14, 30 and 90 Days
Population: The ITT included all participants who were randomized into the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rivaroxaban | Standard-of-care
Number analyzed (Participants) | 51 | 63
Percentage of Participants
  Up to 7 Days | 0 | 0
  Up to 14 Days | 2 | 0
  Up to 30 Days | 3.9 | 1.6
  Up to 90 Days | 3.9 | 6.3

4. Secondary Outcome: Mean Combined Duration of Initial and Subsequent Emergency Department (ED) Hospitalization for Any Reason
Description: Mean combined duration of Initial and subsequent ED Stay and hospitalization for any reason within 30 and 90 days from randomization was analyzed.
Time Frame: Up to 30 and 90 Days
Population: The ITT included all participants who were randomized into the study.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Rivaroxaban | Standard-of-care
Number analyzed (Participants) | 51 | 63
Days
  Within 30 Days | 0.679 (2.0894) | 1.513 (1.9952)
  Within 90 Days | 0.764 (2.1829) | 1.812 (2.714)

5. Secondary Outcome: Treatment Satisfaction Assessment in Participants by Anti-clot Treatment Scale (ACTS)
Description: ACTS is defined as a validated measure for assessing treatment satisfaction. The ACTS comprised of 2 subscales: Burdens (13 items: Item 1 to 13 [how much of limitation from taking part in vigorous physical activities, limitation from usual activities, bothered by bruising, bothered to avoid other medicines, limitation to diet, daily hassle, occasional hassle, difficult to follow treatment, time-consuming, worrying, frustrating, burden, negative impact on life respectively) and Benefits (4 items: Items 14 to 17 for evaluating confidence, reassurance, satisfaction, positive impact respectively) as a result of anti-clot treatment. The treatment experience scores ranged from 'Not at all' to 'Extremely' on a 5-point Likert scale (psychometric rating); higher scores indicate greater satisfaction with treatment.
Time Frame: Day 90
Population: The safety population included all randomized participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban | Standard-of-care
Number analyzed (Participants) | 49 | 63
Percentage of participants
  Item 1: Not at all: number analyzed (Participants) | 45 | 55
  Item 1: Not at all | 51.1 | 61.8
  Item 1: A little: number analyzed (Participants) | 45 | 55
  Item 1: A little | 40 | 21.8
  Item 1: Moderately: number analyzed (Participants) | 45 | 55
  Item 1: Moderately | 6.7 | 10.9
  Item 1: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 1: Quite a bit | 2.2 | 1.8
  Item 1: Extremely: number analyzed (Participants) | 45 | 55
  Item 1: Extremely | 0 | 3.6
  Item 2: Not at all: number analyzed (Participants) | 45 | 55
  Item 2: Not at all | 77.8 | 70.9
  Item 2: A little: number analyzed (Participants) | 45 | 55
  Item 2: A little | 13.3 | 20
  Item 2: Moderately: number analyzed (Participants) | 45 | 55
  Item 2: Moderately | 6.7 | 7.3
  Item 2: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 2: Quite a bit | 2.2 | 0
  Item 2: Extremely: number analyzed (Participants) | 45 | 55
  Item 2: Extremely | 0 | 1.8
  Item 3: Not at all: number analyzed (Participants) | 45 | 55
  Item 3: Not at all | 71.1 | 65.5
  Item 3: A little: number analyzed (Participants) | 45 | 55
  Item 3: A little | 22.2 | 21.8
  Item 3: Moderately: number analyzed (Participants) | 45 | 55
  Item 3: Moderately | 2.2 | 5.5
  Item 3: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 3: Quite a bit | 4.4 | 5.5
  Item 3: Extremely: number analyzed (Participants) | 45 | 55
  Item 3: Extremely | 0 | 1.8
  Item 4: Not at all: number analyzed (Participants) | 45 | 55
  Item 4: Not at all | 60 | 52.7
  Item 4: A little: number analyzed (Participants) | 45 | 55
  Item 4: A little | 33.3 | 20
  Item 4: Moderately: number analyzed (Participants) | 45 | 55
  Item 4: Moderately | 4.4 | 9.1
  Item 4: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 4: Quite a bit | 2.2 | 10.9
  Item 4: Extremely: number analyzed (Participants) | 45 | 55
  Item 4: Extremely | 0 | 7.3
  Item 5: Not at all: number analyzed (Participants) | 45 | 55
  Item 5: Not at all | 80 | 60
  Item 5: A little: number analyzed (Participants) | 45 | 55
  Item 5: A little | 17.8 | 16.4
  Item 5: Moderately: number analyzed (Participants) | 45 | 55
  Item 5: Moderately | 0 | 16.4
  Item 5: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 5: Quite a bit | 2.2 | 7.3
  Item 5: Extremely: number analyzed (Participants) | 45 | 55
  Item 5: Extremely | 0 | 0
  Item 6: Not at all: number analyzed (Participants) | 45 | 55
  Item 6: Not at all | 75.6 | 56.4
  Item 6: A little: number analyzed (Participants) | 45 | 55
  Item 6: A little | 20 | 25.5
  Item 6: Moderately: number analyzed (Participants) | 45 | 55
  Item 6: Moderately | 2.2 | 5.5
  Item 6: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 6: Quite a bit | 2.2 | 12.7
  Item 6: Extremely: number analyzed (Participants) | 45 | 55
  Item 6: Extremely | 0 | 0
  Item 7: Not at all: number analyzed (Participants) | 45 | 55
  Item 7: Not at all | 73.3 | 45.5
  Item 7: A little: number analyzed (Participants) | 45 | 55
  Item 7: A little | 22.2 | 30.9
  Item 7: Moderately: number analyzed (Participants) | 45 | 55
  Item 7: Moderately | 4.4 | 20
  Item 7: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 7: Quite a bit | 0 | 1.8
  Item 7: Extremely: number analyzed (Participants) | 45 | 55
  Item 7: Extremely | 0 | 1.8
  Item 8: Not at all: number analyzed (Participants) | 45 | 55
  Item 8: Not at all | 82.2 | 78.2
  Item 8: A little: number analyzed (Participants) | 45 | 55
  Item 8: A little | 15.6 | 12.7
  Item 8: Moderately: number analyzed (Participants) | 45 | 55
  Item 8: Moderately | 0 | 7.3
  Item 8: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 8: Quite a bit | 2.2 | 1.8
  Item 8: Extremely: number analyzed (Participants) | 45 | 55
  Item 8: Extremely | 0 | 0
  Item 9: Not at all: number analyzed (Participants) | 45 | 55
  Item 9: Not at all | 84.4 | 74.5
  Item 9: A little: number analyzed (Participants) | 45 | 55
  Item 9: A little | 15.6 | 21.8
  Item 9: Moderately: number analyzed (Participants) | 45 | 55
  Item 9: Moderately | 0 | 1.8
  Item 9: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 9: Quite a bit | 0 | 1.8
  Item 9: Extremely: number analyzed (Participants) | 45 | 55
  Item 9: Extremely | 0 | 0
  Item 10: Not at all: number analyzed (Participants) | 45 | 55
  Item 10: Not at all | 48.9 | 43.6
  Item 10: A little: number analyzed (Participants) | 45 | 55
  Item 10: A little | 28.9 | 16.4
  Item 10: Moderately: number analyzed (Participants) | 45 | 55
  Item 10: Moderately | 8.9 | 18.2
  Item 10: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 10: Quite a bit | 11.1 | 10.9
  Item 10: Extremely: number analyzed (Participants) | 45 | 55
  Item 10: Extremely | 2.2 | 10.9
  Item 11: Not at all: number analyzed (Participants) | 45 | 55
  Item 11: Not at all | 77.8 | 60
  Item 11: A little: number analyzed (Participants) | 45 | 55
  Item 11: A little | 17.8 | 16.4
  Item 11: Moderately: number analyzed (Participants) | 45 | 55
  Item 11: Moderately | 4.4 | 7.3
  Item 11: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 11: Quite a bit | 0 | 9.1
  Item 11: Extremely: number analyzed (Participants) | 45 | 55
  Item 11: Extremely | 0 | 7.3
  Item 12: Not at all: number analyzed (Participants) | 45 | 54
  Item 12: Not at all | 84.4 | 64.8
  Item 12: A little: number analyzed (Participants) | 45 | 54
  Item 12: A little | 15.6 | 18.5
  Item 12: Moderately: number analyzed (Participants) | 45 | 54
  Item 12: Moderately | 0 | 9.3
  Item 12: Quite a bit: number analyzed (Participants) | 45 | 54
  Item 12: Quite a bit | 0 | 3.7
  Item 12: Extremely: number analyzed (Participants) | 45 | 54
  Item 12: Extremely | 0 | 3.7
  Item 13: Not at all: number analyzed (Participants) | 45 | 55
  Item 13: Not at all | 64.4 | 54.5
  Item 13: A little: number analyzed (Participants) | 45 | 55
  Item 13: A little | 28.9 | 18.2
  Item 13: Moderately: number analyzed (Participants) | 45 | 55
  Item 13: Moderately | 4.4 | 14.5
  Item 13: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 13: Quite a bit | 2.2 | 7.3
  Item 13: Extremely: number analyzed (Participants) | 45 | 55
  Item 13: Extremely | 0 | 5.5
  Item 14: Not at all: number analyzed (Participants) | 45 | 55
  Item 14: Not at all | 4.4 | 5.5
  Item 14: A little: number analyzed (Participants) | 45 | 55
  Item 14: A little | 8.9 | 7.3
  Item 14: Moderately: number analyzed (Participants) | 45 | 55
  Item 14: Moderately | 20 | 21.8
  Item 14: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 14: Quite a bit | 26.7 | 38.2
  Item 14: Extremely: number analyzed (Participants) | 45 | 55
  Item 14: Extremely | 40 | 27.3
  Item 15: Not at all: number analyzed (Participants) | 45 | 54
  Item 15: Not at all | 4.4 | 5.6
  Item 15: A little: number analyzed (Participants) | 45 | 54
  Item 15: A little | 8.9 | 5.6
  Item 15: Moderately: number analyzed (Participants) | 45 | 54
  Item 15: Moderately | 20 | 24.1
  Item 15: Quite a bit: number analyzed (Participants) | 45 | 54
  Item 15: Quite a bit | 35.6 | 42.6
  Item 15: Extremely: number analyzed (Participants) | 45 | 54
  Item 15: Extremely | 31.1 | 22.2
  Item 16: Not at all: number analyzed (Participants) | 45 | 55
  Item 16: Not at all | 8.9 | 5.5
  Item 16: A little: number analyzed (Participants) | 45 | 55
  Item 16: A little | 2.2 | 9.1
  Item 16: Moderately: number analyzed (Participants) | 45 | 55
  Item 16: Moderately | 15.6 | 9.1
  Item 16: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 16: Quite a bit | 33.3 | 45.5
  Item 16: Extremely: number analyzed (Participants) | 45 | 55
  Item 16: Extremely | 40 | 30.9
  Item 17: Not at all: number analyzed (Participants) | 45 | 55
  Item 17: Not at all | 2.2 | 7.3
  Item 17: A little: number analyzed (Participants) | 45 | 55
  Item 17: A little | 13.3 | 7.3
  Item 17: Moderately: number analyzed (Participants) | 45 | 55
  Item 17: Moderately | 17.8 | 18.2
  Item 17: Quite a bit: number analyzed (Participants) | 45 | 55
  Item 17: Quite a bit | 28.9 | 43.6
  Item 17: Extremely: number analyzed (Participants) | 45 | 55
  Item 17: Extremely | 37.8 | 23.6

6. Secondary Outcome: Percentage of Participants Satisfied Using Site-of-Care Satisfaction Questionnaire
Description: The Satisfaction to Site-of-Care Questionnaire (standard-of-care versus early discharge on rivaroxaban therapy) was administered after 7 days on anticoagulant therapy. Satisfaction to Site-of-Care (hospitalization versus home care) rates the participant's level of satisfaction to care and location with care received as well as preference to location of care provided. Participants rated the 3 items of this scale of 1=Very satisfied; 2=Quite satisfied; 3=Neither; 4=Quite dissatisfied; and 5=Very dissatisfied for satisfaction questions and for the 1 preference question responses included 1=In the hospital; 2=In the community; and 3=No preference. Higher score indicates more level of satisfaction.
Time Frame: Day 7
Population: The safety population included all randomized participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban | Standard-of-care
Number analyzed (Participants) | 49 | 63
Percentage of participants
  Satisfaction level: Very Satisfied: number analyzed (Participants) | 48 | 59
  Satisfaction level: Very Satisfied | 60.4 | 62.7
  Satisfaction level: Quite Satisfied: number analyzed (Participants) | 48 | 59
  Satisfaction level: Quite Satisfied | 33.3 | 23.7
  Satisfaction level: Neither: number analyzed (Participants) | 48 | 59
  Satisfaction level: Neither | 4.2 | 6.8
  Satisfaction level: Quite Dissatisfied: number analyzed (Participants) | 48 | 59
  Satisfaction level: Quite Dissatisfied | 2.1 | 5.1
  Satisfaction level: Very Dissatisfied: number analyzed (Participants) | 48 | 59
  Satisfaction level: Very Dissatisfied | 0 | 1.7
  Location of care: Very Satisfied: number analyzed (Participants) | 48 | 59
  Location of care: Very Satisfied | 62.5 | 59.3
  Location of care: Quite Satisfied: number analyzed (Participants) | 48 | 59
  Location of care: Quite Satisfied | 33.3 | 30.5
  Location of care: Neither: number analyzed (Participants) | 48 | 59
  Location of care: Neither | 4.2 | 6.8
  Location of care: Quite Dissatisfied: number analyzed (Participants) | 48 | 59
  Location of care: Quite Dissatisfied | 0 | 1.7
  Location of care: Very Dissatisfied: number analyzed (Participants) | 48 | 59
  Location of care: Very Dissatisfied | 0 | 1.7
  Preference of care: In the Hospital: number analyzed (Participants) | 48 | 59
  Preference of care: In the Hospital | 18.8 | 47.5
  Preference of care: In the Community: number analyzed (Participants) | 48 | 59
  Preference of care: In the Community | 50 | 40.7
  Preference of care: No Preference: number analyzed (Participants) | 48 | 59
  Preference of care: No Preference | 31.3 | 11.9

ADVERSE EVENTS:
Time Frame: Approximately 2.5 years
Description: The safety population included all randomized participants who took at least 1 dose of study drug.
Arm/Group | Rivaroxaban | Standard-of-care
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/63
Serious Adverse Events (participants affected / at risk) | 5/49 | 7/63
Other Adverse Events (participants affected / at risk) | 15/49 | 13/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (N=49) | Standard-of-care (N=63)
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Systemic Inflammatory Response Syndrome (General disorders) | 0 | 1
Device Related Infection (Infections and infestations) | 1 | 0
Embolic Pneumonia (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
May-Thurner Syndrome (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (N=49) | Standard-of-care (N=63)
Chest Pain (General disorders) | 5 | 3
Non-Cardiac Chest Pain (General disorders) | 0 | 2
Sinusitis (Infections and infestations) | 2 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Headache (Nervous system disorders) | 2 | 3
Menorrhagia (Reproductive system and breast disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2015-06-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT02584660/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT02584660/SAP_001.pdf